CLINICAL TRIAL: NCT06104150
Title: Transporte Eritrocitario de Lactato en Ejercicio
Brief Title: Erythrocyte Transport of Lactate During Exercise (TELE Project)
Acronym: TELE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Madrid (Other)
Responsible Party: Principal Investigator, Rocío Cupeiro, PhD, Physical Activity and Sports PhD (Associate Professor), Technical University of Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PINV-18-ENW9ML-92-B2287R
Record Dates: First submitted 2023-10-19; First posted 2023-10-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Energy Metabolism
Keywords: lactate kinetics; MCT1; erythrocyte lactate; T1470A polymorphism; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervallic submaximal test (Experimental): Intervallic exercise test
  Interventions: Other: Intervallic submaximal exercise test

INTERVENTIONS:
Other: Intervallic submaximal exercise test — Intervallic submáximal exercise test on a cycle ergometer: 5 min warm-up at 80% of First Lactate Threshold (LT1), and subsequent sets of 1.5 min at 20% above the Second Lactate Threshold (LT2) alternated with recoveries of 5 min at 80% of LT1, ending with a 20 min recovery at 80% of LT1.
  Other Names: Interval exercise training

SUMMARY:
The goals of this clinical trial are:

1. to study lactate kinetic between plasma and erythrocytes during an intervallic exercise and its subsequent recovery, considering the blood pH, the genotype for the T1470A polymorphism of the SLC16A1 gene (rs1049434), and the amount of MCT1 in erythrocytes membrane;
2. to analyze the levels of MCT1 in the erythrocytes membrane according to training status and genotype for the T1470A polymorphism of SLC16A1 (rs1049434).

For this, the project will have two phases:

* In phase I, trained participants will perform one maximal incremental test and one intervallic submaximal test with a final active recovery.
* Phase II, levels of the MCT1 protein in the erythrocyte membrane will be quantified from trained and sedentary participants.

DETAILED DESCRIPTION:
Introduction

Lactate is the end product of glycolysis and has the capacity to be transported from one cell to another, performing numerous functions. This transport is mainly through several monocarboxylate transporters (MCT). The most predominant is MCT1, which transfers lactate bidirectionally depending on the lactate concentration and pH on each side of the membrane. MCT1 is ubiquitous, being present in most human tissues like the erythrocyte membrane, indicating that these cells are capable of carrying lactate throughout the bloodstream. Some studies have described lactate kinetics between the different blood compartments (erythrocyte-plasma) during incremental and steady-state exercises, but not during intermittent exercise and/or recovery after exercise. Moreover, several studies have observed that the function of MCT1 is conditioned by the presence of a genetic variant: the T1470A polymorphism (rs1049434), which involves a substitution of aspartic acid for glutamic acid at position 490 of the protein. Data suggest that an AA (Glu/Glu) genotype for this single nucleotide polymorphism (or SNP) leads to a higher lactate transport capacity than the TT (Arg/Arg) profile. However, no study has analyzed if this SNP directly affects erythrocyte MCT1 function or content Therefore, the two general objectives of this clinical trial are:

1. to study lactate kinetic between plasma and erythrocytes during an intervallic exercise and its subsequent recovery, considering the blood pH, the genotype for the T1470A polymorphism of the SLC16A1 gene (rs1049434), and the amount of MCT1 in erythrocytes membrane;
2. to analyze the levels of MCT1 in the erythrocytes membrane according to training status and genotype for the T1470A polymorphism of SLC16A1 (rs1049434).

Procedures

The study will be divided into two phases, each of which will be primarily oriented toward achieving one of two general objectives:

* Phase I: Focused primarily on the study of lactate kinetics between blood compartments during exercise.
* Phase II: Focused primarily on the analysis of the amount of MCT1 in the erythrocyte membrane.

For both phases, volunteers will be informed and sign an informed consent form before a blood sample is taken for genotyping. Once the genotype is known, only those participants with AA or TT genotype will be selected.

The tests that will be performed throughout Phase I will be the following:

* Once participants with the genotypes AA and TT are selected, they will perform a step incremental test until exhaustion to determine the first and second lactate threshold. These thresholds will be determined by measuring lactate concentration from capillary blood samples from the earlobe.
* Finally, an intervallic exercise protocol will be performed starting with 1 min rest followed by a 5 min warm up at an intensity equal to 80% of the first lactate threshold. This is followed by 4 sets of 1 min 30 sec at an intensity 20% above the second lactate threshold, with recovery intervals of 5 min at 80% of the first lactate threshold. After the 4 sets, a final recovery of 20 min at 80% of the first lactate threshold will be performed. During this test, capillary blood samples from the earlobe and venous blood samples from the forearm will be analyzed for lactate concentration.

The procedure for the Phase II will be the following:

* Once participants with the genotype AA and TT are selected, venous blood will be extracted from their forearm at rest.
* Physical activity levels from all the participants will be quantified using the International Physical Activity Questionnaire (IPAQ).
* Analysis of the erythrocyte MCT1 protein content by flow cytometry will be performed from the venous blood samples.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 25 kg/m2
* Not smoker
* In the case of trained participants: training at least 5 hours/week, of which at least 3 must be aerobic/anaerobic endurance training. Presentation of a medical certificate attesting to their medical fitness (capability) to perform intense physical exercise.
* In the case of sedentary participants, less than 1 day of training per week or less than 2 hours of structured exercise per week.

Exclusion Criteria:

* Presenting any pathology that could impede the correct performance of the tests, or could influence the main study variables.
* In the case of the female sample, having irregular menstrual cycles, oligomenorrhea or amenorrhea.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Plasma-Erythrocyte lactate difference | Through Phase I of the project, only in the intervallic submaximal test. Average of 3 years
  Difference between lactate concentration inside the erythrocytes and lactate concentration in plasma, expressed in mMol/L (Millimoles Per Liter), from venous blood extracted during the intervallic test from the antecubital vein.
Level of Monocarboxylate Transporter 1 in erythrocytes membrane | Through study completion, average of 5 years, an average of 2 months per participant
  Protein abundance of the monocarboxylate transporter 1 in erythrocyte membranes. It is measured using flow cytometry, from venous blood extracted from the forearm in rest state.

SECONDARY OUTCOMES:
Erythrocyte lactate concentration | Through Phase I of the project, only in the intervallic submaximal test. Average of 3 years
  Lactate concentration inside the erythrocytes, expressed in mMol/L (Millimoles Per Liter), measured in erythrocytes extracted from processed venous blood.
  Lactate concentration is measured in the supernatant obtained after the lysis and centrifugation of the solid part of the blood (mainly erythrocytes), separated by centrifugation. Venous blood samples are extracted during the intervallic test from the antecubital vein.
Plasma lactate concentration | Through Phase I of the project, only in the intervallic submaximal test. Average of 3 years
  Lactate concentration, expressed in mMol/L (Millimoles Per Liter), measured in the plasma of centrifugated venous blood, using a lactate analyzer.
  Lactate concentration is measured in the plasma obtained from venous blood extracted during the intervallic test from the antecubital vein.
Blood lactate concentration | Through Phase I of the project, only in the intervallic submaximal test. Average of 3 years
  Lactate concentration, expressed in mMol/L (Millimoles Per Liter), measured from whole venous blood extracted during the intervallic test from the antecubital vein.
Blood pH | Through Phase I of the project, only in the intervallic submaximal test. Average of 3 years
  Level of blood pH measured in venous blood extracted during the intervallic test from the antecubital vein.

OTHER OUTCOMES:
Genotype for the rs1049434 polymorphism of the SLC16A1 (MCT1) gene | Through sample recruitment, average of 5 years, an average of 1 month per participant
  Genotype for the Asp490Glu (T1470A) (rs1049434) polymorphism of the SLC16A1 (MCT1) gene, resulting in one of the following three profiles: TT (Arg/Arg), TA (Arg/Glu) or AA (Glu/Glu)
Physical Activity level | Through sample recruitment, average of 5 years, an average of 1 month per participant
  The IPAQ self-reported questionnaire will be used to quantify physical activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Cupeiro, PhD, Principal Investigator — Universidad Politecnica de Madrid
Locations (2):
- Spain (2):
  - Laboratorio de Pediatría. School of Medicine. Univesidad de Cantabria, Santander, Cantabria
  - Laboratorio de Fisiología del Esfuerzo. Facultad de Ciencias de la Actividad Física y del Deporte (INEF). Universidad Politécnica de Madrid, Madrid, Madrid

REFERENCES:
- [Derived] Benitez-Munoz JA, Rojo-Tirado MA, Benito Peinado PJ, Murias JM, Gonzalez-Lamuno D, Cupeiro R. Greater Relative First and Second Lactate Thresholds in Females Compared With Males: Consideration for Exercise Prescription. Int J Sports Physiol Perform. 2024 Oct 28;20(1):30-36. doi: 10.1123/ijspp.2024-0079. Print 2025 Jan 1. PMID 39467538